CLINICAL TRIAL: NCT03051971
Title: A Pilot Study of Medicated Aerosol Delivery Using A Jet Nebulizer Versus A Vibrating Mesh Nebulizer in COPD Exacerbation
Brief Title: Medicated Aerosol Delivery Using A Jet Nebulizer Versus A Vibrating Mesh Nebulizer in COPD Exacerbation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was abandoned.
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-281
Record Dates: First submitted 2017-01-30; First posted 2017-02-14 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Jet nebulizer (Active Comparator): short-acting bronchodilator (albuterol and/or ipratropium bromide) according to standard of care practices and physician discretion will be administered with a jet nebulizer
  Interventions: Device: Jet Nebulizer
- Vibrating Mesh Nebulizer (Active Comparator): short-acting bronchodilator (albuterol and/or ipratropium bromide) according to standard of care practices and physician discretion will be administered with a vibrating mesh nebulizer
  Interventions: Device: Vibrating Mesh Nebulizer

INTERVENTIONS:
Device: Vibrating Mesh Nebulizer — short-acting bronchodilator medication delivered with a vibrating mesh nebulizer via mouthpiece, valved facemask or non-invasive ventilation mask
  Other Names: Aergoen Ultra nebulizer
  Arms: Vibrating Mesh Nebulizer
Device: Jet Nebulizer — short-acting bronchodilator medication delivered with a jet nebulizer via mouthpiece, valved facemask or non-invasive ventilation mask
  Other Names: MistyFast nebulizer
  Arms: Jet nebulizer

SUMMARY:
Delivery of inhaled short-acting bronchodilators (SABD) is standard of care in the emergency department (ED) for exacerbation of COPD, the goal of such being rapid reversal of airflow obstruction. However, current guidelines for the delivery of SABDs in spontaneously breathing patients make no distinction whether these medications should be delivered via metered dose inhaler (MDI) or jet nebulizer (JN), the specific medication delivery device having no significant effect on hospital admission or reversal of flow obstruction. However, advancements in nebulizer design, namely FDA-approved vibrating mesh technology, have demonstrated significant improvements relative to JNs and metered dose inhalers in efficiency and amount of drug delivered in in vivo and in vitro studies. Currently there are no clinical trials comparing the use of vibrating mesh nebulizers (VMN) to JNs and their effect on clinically important outcomes. This prospective randomized controlled pilot trial seeks to determine if there are differences in hospital admission due to COPD when a vibrating mesh nebulizer is used versus a jet nebulizer.

DETAILED DESCRIPTION:
Patients ordered to receive a SABD, will be screened for presence of moderate to severe COPD exacerbation; spontaneously breathing patients as well those supported with non-invasive ventilation (NIV) will be screened for inclusion.

Upon consent, the patient will be randomized to receive the ordered SABD via a JN (MistyFast, Carefusion-BD, CA) or VMN (Aerogen Ultra, Aerogen, Galway, Ireland).

Included subjects will receive therapy with a mouthpiece interface. In the case a patient is unable to tolerate, maintain a tight seal around the mouthpiece or otherwise not perform aerosol therapy with a mouthpiece, a valved-aerosol mask (I-Guard aerosol mask, Salter Labs, Lake Forest, IL) will be utilized.

Subjects that require NIV, whether on admission to the ED or in the face of escalating therapy, will receive NIV via a non-vented, oronasal mask and the allocated nebulizer will be placed distal to the leak in the NIV circuit (between the mask and circuit). Patients will receive positive expiratory and/or inspiratory pressure at specific settings determined by the prescribing physician and clinical team.

Subjects will be re-evaluated and clinical data collected following delivery of the initial SABD treatment that includes signs of possible side effects.

The prescribing physician and clinical team will determine the need for additional SABD therapy beyond the initial therapy. Subjects indicated and ordered for additional administration of SABD will continue to receive SABD with the randomly allocated aerosol delivery device. Subjects will be re-evaluated and assessed for possible side effects after delivery of the additional SABD.

The initial order, as well as all subsequent orders for SABD medication will be at the discretion of the physician and clinical team. The type and dosage of medication and the approximate timing of medication delivery designated in the study protocol is according to and correlates with the standard practices. The process of determining need by the clinical team and administering additional SABD, followed by evaluation, will continue up to a total of four SABD treatments. If at any point following a SABD treatment, the clinical team assesses the subject and determines that no additional therapy is indicated, the subject will not receive additional SABD. Clinical data will be collected following each SABD administered (approximately every 30 minutes) and conclude at 120 min after randomization.

Subjects requiring the need for endotracheal intubation and mechanical ventilator support, immediate or in escalation of support, will be at the discretion of the attending physician. Subjects requiring endotracheal intubation as escalation of therapy following study enrollment will be included in the study analysis. Those subjects requiring the immediate need for endotracheal intubation prior to randomization will be excluded from the study.

Individualized decision regarding hospitalization or discharge to home will be according to the attending physician. Subjects admitted to the hospital for continued inpatient care will continue to receive nebulized bronchodilator therapy, as indicated and ordered, with an aerosol delivery device according to the MWHC bronchodilator protocol and standard practices.

ELIGIBILITY:
Inclusion Criteria:

i. Patients ordered to receive short-acting bronchodilator therapy ii. Patients ≥ 40 years of age iii. Patients with a self-reported history of COPD and/or patients with diagnosed/suspected COPD iv. Patients whose FEV1 is ≤ 50% of predicted or are unable to perform FEV1 maneuver because of airflow-associated respiratory distress or NIV use

Exclusion Criteria:

i. Patients whose indication for SABD therapy is for a clinical indication other than COPD ii. The immediate need for intubation iii. Pregnant women iv. Non-English speakers

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | through study completion (approx 1 year)
  hospitalization rate among COPD exacerbation patients in the ED receiving SABD via jet nebulizer versus those receiving SABD via VMN

SECONDARY OUTCOMES:
ICU admission | through study completion (approx 1 year)
  Percent of patients with COPD exacerbation treated with SABD via VMN versus JN admitted to an intensive care environment
Hospital length of stay | through study completion (approx 1 year)
  Hospital length of stay for patients with COPD exacerbation treated with SABD via VMN versus JN
NIV in escalation of respiratory support | through study completion (approx 1 year)
  Percentage of patients with COPD exacerbation treated with SABD via VMN versus JN that require NIV in escalation of respiratory support
Duration of NIV support | through study completion (approx 1 year)
  Duration of NIV support in patients with COPD exacerbation treated with SABD via VMN versus JN
Intubation in escalation of respiratory support | through study completion (approx 1 year)
  Percentage of patients with COPD exacerbation treated with SABD via VMN versus JN that require intubation in escalation of respiratory support
Percentage change in FEV1 | through study completion (approx 1 year)
  Percentage change in FEV1 in patients with COPD exacerbation treated with SABD via VMN versus JN
Amount of short-acting bronchodilator medication | through study completion (approx 1 year)
  The amount of SABD aerosol therapy administered to patients with COPD exacerbation treated with SABD via VMN versus JN
Hospital readmission within 30 days | through study completion (approx 1 year)
  Percentage of patients treated with SABD via VMN versus JN that are readmitted to the hospital within thirty days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Kriner, RRT, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No